CLINICAL TRIAL: NCT07378605
Title: Effect of Intraoperative Salbutamol Administration on Mechanical Power and Respiratory Mechanics in Obese Patients Undergoing Laparoscopic Bariatric Surgery
Acronym: Bariatric
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Saglik Bilimleri Universitesi Gazi Yasargil Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Hülya Tosun Söner, Saglik Bilimleri Universitesi Gazi Yasargil Training and Research Hospital, Saglik Bilimleri Universitesi Gazi Yasargil Training and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: Hts
Record Dates: First submitted 2025-12-26; First posted 2026-01-30 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Bariatric Surgery
MeSH Terms: interventions — Albuterol; Saline Solution; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Salbutamol Group (Experimental): Participants in this arm will receive intraoperative salbutamol administration in addition to standard general anesthesia and mechanical ventilation during laparoscopic bariatric surgery.
  Interventions: Drug: Salbutamol (Ventolin®)
- Control Group (Placebo Comparator): Participants in this arm will receive intraoperative administration of normal saline (0.9% sodium chloride) via the respiratory circuit, in addition to standard general anesthesia and mechanical ventilation during laparoscopic bariatric surgery.
  Interventions: Drug: Normal Saline (0.9% Sodium Chloride)

INTERVENTIONS:
Drug: Salbutamol (Ventolin®) — Salbutamol will be administered intraoperatively via the respiratory circuit during mechanical ventilation to assess its effect on mechanical power and respiratory mechanics.
  Arms: Salbutamol Group
Drug: Normal Saline (0.9% Sodium Chloride) — Normal saline will be administered intraoperatively via the respiratory circuit in the same volume and manner as salbutamol to serve as a placebo
  Arms: Control Group

SUMMARY:
The primary objective of this study is to evaluate the effect of intraoperative salbutamol administration on mechanical power in obese patients undergoing laparoscopic bariatric surgery under general anesthesia. Mechanical power will be measured at predefined intraoperative time points (T0, T1, and T2), and changes over time will be compared to determine the impact of salbutamol on the overall energy delivered to the respiratory system during mechanical ventilation.

Secondary objectives include the assessment of intraoperative respiratory mechanics, including peak airway pressure (Ppeak), plateau pressure (Pplat), driving pressure (Pdrive), airway resistance (Raw), and lung compliance, as well as gas exchange parameters (SpO₂, EtCO₂) and hemodynamic variables (mean arterial pressure). Postoperative pulmonary outcomes will be evaluated using the Melbourne Group Scale (MGS), with a score greater than 4 indicating the presence of postoperative pulmonary complications. The study aims to investigate whether improvement in intraoperative mechanical power and respiratory mechanics is associated with a reduction in postoperative pulmonary complications in this high-risk population.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18-65 years

BMI ≥35 kg/m² (candidates for obesity surgery)

Scheduled for elective laparoscopic bariatric surgery

ASA physical status I-III

Signed informed consent

Exclusion Criteria:

Known allergy or contraindication to salbutamol

Severe cardiovascular disease (e.g., recent MI, uncontrolled arrhythmia)

Pre-existing severe pulmonary disease (e.g., severe COPD, asthma exacerbation)

Pregnancy or lactation

Emergency surgery

Use of β-agonists or bronchodilators within 24 hours prior to surgery

Patients with inability to provide informed consent

-

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-03-15 (Estimated)

PRIMARY OUTCOMES:
Change in intraoperative mechanical power | Baseline (intraoperative, after establishment of pneumoperitoneum and before Ventolin or saline administration)
  Mechanical power will be measured directly by the ventilator/respiratory monitoring device using ventilator parameters (tidal volume, respiratory rate, peak and plateau pressures, driving pressure, and compliance) at T0, T1, and T2. The primary outcome is the difference in mechanical power between the Salbutamol and placebo groups over time.

SECONDARY OUTCOMES:
Peak airway pressure (Ppeak) | Baseline (intraoperative, after establishment of pneumoperitoneum and before Ventolin or saline administration)
  Peak airway pressure will be measured directly by the ventilator/respiratory monitoring device at T0, T1, and T2 to assess intraoperative respiratory mechanics.
Plateau pressure (Pplat) | Baseline (intraoperative, after establishment of pneumoperitoneum and before Ventolin or saline administration)
  Plateau pressure will be measured by the ventilator device at T0, T1, and T2 to evaluate changes in lung mechanics.
Driving pressure (Pdrive) | Baseline (intraoperative, after establishment of pneumoperitoneum and before Ventolin or saline administration)
  Driving pressure (Pplat minus PEEP) will be measured via the ventilator device at all intraoperative time points to assess lung stress.
Airway resistance (Raw) | Baseline (intraoperative, after establishment of pneumoperitoneum and before Ventolin or saline administration)
  Airway resistance will be recorded from the ventilator/monitoring device at each time point to evaluate intraoperative airway changes.
Lung compliance | Baseline (intraoperative, after establishment of pneumoperitoneum and before Ventolin or saline administration)
  Lung compliance will be measured by the ventilator at T0, T1, and T2 to assess changes in respiratory mechanics.
Lung elastance (E) | Baseline (intraoperative, after establishment of pneumoperitoneum and before Ventolin or saline administration)
  Lung elastance will be measured directly by the ventilator/monitoring device at each intraoperative time point (T0, T1, T2) to evaluate the stiffness of the respiratory system and its changes due to pneumoperitoneum and Ventolin/SF administration.
Heart rate (HR / Nabız) | Baseline (intraoperative, after establishment of pneumoperitoneum and before Ventolin or saline administration)
  Heart rate will be monitored continuously and recorded at T0, T1, and T2 to evaluate intraoperative hemodynamic stability and potential effects of pneumoperitoneum and Ventolin/SF administration.
Mean arterial pressure (MAP) | Baseline (intraoperative, after establishment of pneumoperitoneum and before Ventolin or saline administration)
  Mean arterial pressure will be monitored continuously and recorded at T0, T1, and T2 to assess intraoperative hemodynamic stability and the effects of pneumoperitoneum and Ventolin/SF administration.
Postoperative pulmonary complications (Melbourne Group Scale >4) | First assessment: Within 24 hours postoperatively Second assessment: 48 hours postoperatively Third assessment: Immediately before hospital discharge
  Incidence of postoperative pulmonary complications will be assessed using the Melbourne Group Scale (MGS). A score greater than 4 indicates the presence of a postoperative pulmonary complication. Criteria include:
  Temperature >38°C
  White cell count >11.2 ×10⁹/L or use of respiratory antibiotics
  Physician diagnosis of pneumonia or chest infection
  Chest X-ray findings of atelectasis or consolidation
  Production of purulent (yellow/green) sputum different from preoperative sputum
  Positive microbiological analysis of sputum
  SpO₂ <90% in ambient air
  Re-admission to or prolonged stay (>36 h) in ICU/high dependency unit for respiratory problems
  Patients meeting ≥4 of these criteria at any assessment point will be recorded as having a postoperative pulmonary complication.

CONTACTS AND LOCATIONS:
Locations (1):
- Health Sciences University Gazi Yaşargil Training and Research Hospital, Kayapınar, Diyarbakır, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No